CLINICAL TRIAL: NCT02062593
Title: Defining a Gold Standard for Ischaemia: Effects of Interventional Revascularisation Versus Optimum Medical Therapy on Exercise Capacity in Patients With Stable Coronary Artery Disease
Brief Title: Objective Randomised Blinded Investigation With Optimal Medical Therapy of Angioplasty in Stable Angina
Acronym: ORBITA
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Imperial College London (Other)
Collaborators: Volcano Corporation (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: ORBITA-1
Record Dates: First submitted 2014-01-31; First posted 2014-02-13 (Estimated); Results first posted 2021-04-22 (Actual); Last update posted 2024-01-22 (Actual); Status verified 2024-01

CONDITIONS: Stable Angina
Keywords: Stable angina; Percutaneous coronary intervention; Optimal medical therapy; Sham-control
MeSH Terms: conditions — Angina, Stable | interventions — Angioplasty, Balloon; Percutaneous Coronary Intervention

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Coronary angioplasty and optimum medical therapy (Active Comparator): Percutaneous coronary intervention and optimal medical therapy
  Interventions: Procedure: Coronary angioplasty
- Sham procedure and optimum medical therapy (Placebo Comparator): Placebo percutaneous coronary intervention and optimal medical therapy with risk factor modification and anti-anginal therapy
  Interventions: Procedure: Coronary angioplasty

INTERVENTIONS:
Procedure: Coronary angioplasty — Percutaneous coronary intervention with drug-eluting stents and modern techniques
  Other Names: Percutaneous coronary intervention

SUMMARY:
In this study the investigators will use careful scientific blinding of patient and their subsequent healthcare staff so that the investigators can determine exactly how much difference coronary angioplasty makes to symptoms and blood supply to the heart. After the 6 weeks blinded phase, all patients will be unblinded and the patients who had undergone sham procedure will be offered the active therapy.

DETAILED DESCRIPTION:
The investigators will perform a multi-centre prospective randomised double-blinded comparison of the treatment of stable angina with percutaneous coronary intervention (PCI) and optimal medical therapy (OMT) versus a sham procedure and OMT. Two hundred patients with stable angina and one or more angiographically significant coronary stenosis of 70% or more in a single vessel that is suitable for angioplasty will be recruited. Baseline investigation of functional capacity and myocardial ischaemic burden will be performed. This will be followed by a coronary angiogram and invasive physiological investigation followed by randomisation to PCI or a sham procedure. Follow-up investigation of functional capacity and myocardial ischaemic burden at 6 weeks will then be performed.

ELIGIBILITY:
Inclusion Criteria:

* Stable angina and at least 1 lesion with angiographic stenosis ≥70% in a single vessel suitable for stent implantation

Exclusion Criteria:

* Acute coronary syndrome
* Previous coronary artery bypass graft surgery
* Left main stem disease
* Contraindications to PCI or drug-eluting stent (DES) implantation
* Heavily calcified or tortuous vessels
* Chronic total occlusion in target vessel
* Life expectancy <2yr
* Pregnancy
* Age <18yr or >85yr
* Angiographic stenosis ≥ 50% in non-target vessel
* Inability to consent

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 230 (Actual)
Dates: Start 2013-12 (Actual); Primary Completion 2017-08 (Actual); Study Completion 2017-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Justin E Davies, MRCP, PhD, Principal Investigator — Imperial College London; Darrel P Francis, MRCP, MD, Study Chair — Imperial College London; Rasha K Al-Lamee, MRCP, Study Director — Imperial College London
Locations (5):
- United Kingdom (5):
  - East Sussex Healthcare NHS Trust, Saint Leonards-on-Sea, East Sussex
  - Basildon and Thurrock University Hospitals NHS Trust, Basildon
  - The Royal Bournemouth and Christchurch Hospitals NHS Trust, Bournemouth
  - Royal Devon & Exeter Foundation Trust, Exeter
  - Imperial College Healthcare NHS Trust, London

REFERENCES:
- [Result] Al-Lamee R, Thompson D, Dehbi HM, Sen S, Tang K, Davies J, Keeble T, Mielewczik M, Kaprielian R, Malik IS, Nijjer SS, Petraco R, Cook C, Ahmad Y, Howard J, Baker C, Sharp A, Gerber R, Talwar S, Assomull R, Mayet J, Wensel R, Collier D, Shun-Shin M, Thom SA, Davies JE, Francis DP; ORBITA investigators. Percutaneous coronary intervention in stable angina (ORBITA): a double-blind, randomised controlled trial. Lancet. 2018 Jan 6;391(10115):31-40. doi: 10.1016/S0140-6736(17)32714-9. Epub 2017 Nov 2. PMID 29103656
- [Derived] Rajkumar CA, Wereski R, Parsonage W, Cullen L, Khamis R, Foley M, Harrell FE Jr, Shun-Shin MJ, Mills NL, Al-Lamee RK. Association Between High-Sensitivity Cardiac Troponin, Myocardial Ischemia, and Revascularization in Stable Coronary Artery Disease. J Am Coll Cardiol. 2022 May 31;79(21):2185-2187. doi: 10.1016/j.jacc.2022.03.369. No abstract available. PMID 35618353
- [Derived] Rajkumar CA, Shun-Shin M, Seligman H, Ahmad Y, Warisawa T, Cook CM, Howard JP, Ganesananthan S, Amarin L, Khan C, Ahmed A, Nowbar A, Foley M, Assomull R, Keenan NG, Sehmi J, Keeble TR, Davies JR, Tang KH, Gerber R, Cole G, O'Kane P, Sharp ASP, Khamis R, Kanaganayagam G, Petraco R, Ruparelia N, Malik IS, Nijjer S, Sen S, Francis DP, Al-Lamee R. Placebo-Controlled Efficacy of Percutaneous Coronary Intervention for Focal and Diffuse Patterns of Stable Coronary Artery Disease. Circ Cardiovasc Interv. 2021 Aug;14(8):e009891. doi: 10.1161/CIRCINTERVENTIONS.120.009891. Epub 2021 Aug 3. PMID 34340523
- [Derived] McCreanor V, Nowbar A, Rajkumar C, Barnett AG, Francis D, Graves N, Boden WE, Weintraub WS, Al-Lamee R, Parsonage WA. Cost-effectiveness analysis of percutaneous coronary intervention for single-vessel coronary artery disease: an economic evaluation of the ORBITA trial. BMJ Open. 2021 Feb 9;11(2):e044054. doi: 10.1136/bmjopen-2020-044054. PMID 33563623
- [Derived] Foley M, Rajkumar CA, Shun-Shin M, Ganesananthan S, Seligman H, Howard J, Nowbar AN, Keeble TR, Davies JR, Tang KH, Gerber R, O'Kane P, Sharp ASP, Petraco R, Malik IS, Nijjer S, Sen S, Francis DP, Al-Lamee R. Achieving Optimal Medical Therapy: Insights From the ORBITA Trial. J Am Heart Assoc. 2021 Feb 2;10(3):e017381. doi: 10.1161/JAHA.120.017381. Epub 2021 Jan 26. PMID 33496201
- [Derived] Al-Lamee RK, Shun-Shin MJ, Howard JP, Nowbar AN, Rajkumar C, Thompson D, Sen S, Nijjer S, Petraco R, Davies J, Keeble T, Tang K, Malik I, Bual N, Cook C, Ahmad Y, Seligman H, Sharp ASP, Gerber R, Talwar S, Assomull R, Cole G, Keenan NG, Kanaganayagam G, Sehmi J, Wensel R, Harrell FE Jr, Mayet J, Thom S, Davies JE, Francis DP. Dobutamine Stress Echocardiography Ischemia as a Predictor of the Placebo-Controlled Efficacy of Percutaneous Coronary Intervention in Stable Coronary Artery Disease: The Stress Echocardiography-Stratified Analysis of ORBITA. Circulation. 2019 Dec 10;140(24):1971-1980. doi: 10.1161/CIRCULATIONAHA.119.042918. Epub 2019 Nov 11. PMID 31707827
- [Derived] Al-Lamee R, Howard JP, Shun-Shin MJ, Thompson D, Dehbi HM, Sen S, Nijjer S, Petraco R, Davies J, Keeble T, Tang K, Malik IS, Cook C, Ahmad Y, Sharp ASP, Gerber R, Baker C, Kaprielian R, Talwar S, Assomull R, Cole G, Keenan NG, Kanaganayagam G, Sehmi J, Wensel R, Harrell FE, Mayet J, Thom SA, Davies JE, Francis DP. Fractional Flow Reserve and Instantaneous Wave-Free Ratio as Predictors of the Placebo-Controlled Response to Percutaneous Coronary Intervention in Stable Single-Vessel Coronary Artery Disease. Circulation. 2018 Oct 23;138(17):1780-1792. doi: 10.1161/CIRCULATIONAHA.118.033801. PMID 29789302

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Coronary Angioplasty and Optimum Medical Therapy | Sham Procedure and Optimum Medical Therapy
Started | 105 | 95
Completed | 105 | 91
Not Completed | 0 | 4

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Coronary Angioplasty and Optimum Medical Therapy | Sham Procedure and Optimum Medical Therapy | Total
Number analyzed (Participants) | 105 | 95 | 200
Age, Continuous [Mean (Standard Deviation); unit: years] | 65.9 (9.5) | 66.1 (8.4) | 66 (9)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 31 | 23 | 54
  Male | 74 | 72 | 146
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Number; unit: participants]
  United Kingdom | 105 | 95 | 200

OUTCOME MEASURES:

1. Primary Outcome: Exercise Time on Treadmill
Description: Measured in seconds on Modified Bruce exercise treadmill protocol
Time Frame: 6 weeks
Population: No exercise time data available for 1 patient in PCI group and 5 patients in placebo group.
Measure: Mean (95% Confidence Interval); unit: seconds
Arm/Group | Coronary Angioplasty and Optimum Medical Therapy | Sham Procedure and Optimum Medical Therapy
Number analyzed (Participants) | 104 | 90
seconds | 28.4 [11.6 to 45.1] | 11.8 [-7.8 to 31.3]

ADVERSE EVENTS:
Time Frame: Total study time 12 weeks
Arm/Group | Coronary Angioplasty and Optimum Medical Therapy | Sham Procedure and Optimum Medical Therapy
All-Cause Mortality (participants affected / at risk) | 0/105 | 0/95
Serious Adverse Events (participants affected / at risk) | 4/105 | 14/95
Other Adverse Events (participants affected / at risk) | 0/105 | 0/95
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Coronary Angioplasty and Optimum Medical Therapy (N=105) | Sham Procedure and Optimum Medical Therapy (N=95)
Major bleeding (Blood and lymphatic system disorders) | 2 (2) | 3 (3)
Acute confusion (Nervous system disorders) | 1 (1) | 0 (0)
Crossover to PCI (Cardiac disorders) | 0 (0) | 4 (4)
Wire snapped required snare retrieval (Cardiac disorders) | 1 (1) | 0 (0)
Pulmonary oedema (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 2 (2)
Acute coronary syndrome (Cardiac disorders) | 0 (0) | 1 (1)
Hospitalisation for atypical chest pain (Cardiac disorders) | 0 (0) | 1 (1)
Hospitalisation for right heart failure (Cardiac disorders) | 0 (0) | 1 (1)
Hospitalisation for leg pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Severe drug reaction (Immune system disorders) | 0 (0) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2014-08-14): https://cdn.clinicaltrials.gov/large-docs/93/NCT02062593/Prot_SAP_000.pdf